CLINICAL TRIAL: NCT00272831
Title: A Randomised, Double-Blind, Placebo-Controlled Study of Cilostazol 100 mg Twice Daily in the Treatment of Diabetic Nephropathy in Hong Kong Chinese
Brief Title: The Use of Cilostazol in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr Peter CY Tong, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PWH 2005-146-T
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Diabetic nephropathy; Macroalbuminuria; Pletaal
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Nephropathies | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Active Comparator): Cilostazol 100 mg twice daily
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100 mg twice daily
  Other Names: Pletaal
  Arms: Cilostazol
Drug: Placebo — 1 tablet twice daily
  Arms: Placebo

SUMMARY:
Patients with type 2 diabetes have a long duration of disease for the development of complications. Among all complications, microangiopathic complications are major causes of mortality and morbidity in diabetic patients. In Asia, patients with type 2 diabetes are particularly susceptible to the development of kidney disease. Patients with diabetic kidney disease have more adverse metabolic profiles and increased risk of having other complications such as blindness, stroke, heart attack and nerve damage than those without. Despite receiving the best of care, the combined event rate of death, cardiovascular disease and end stage kidney disease in diabetic patients with renal impairment remained as high as 10% per year.

Cilostazol reduces platelet aggregation and prevents formation of blood clots. Furthermore, cilostazol treatment has been shown to reduce serum triglyceride concentrations and increase HDL-cholesterol levels. In this randomized placebo-controlled, double-blinded study, the investigators hypothesize that Cilostazol may reduce the rate of decline in renal function in Chinese patients with type 2 diabetes and mild to moderate renal impairment. Sixty patients will be randomised to receive either Cilostazol 100 mg twice daily or placebo for 12 months. The effect of Cilostazol on the progression of diabetic nephropathy, as defined by rates of decline in glomerular filtration rate, serum creatinine and urinary albumin excretion rate will be measured. The results will provide additional insight on the management of diabetic kidney disease which is prevalent among Chinese diabetic patients in Hong Kong.

DETAILED DESCRIPTION:
Hypothesis:

Cilostazol reduces the rate of decline in renal function in Chinese patients with type 2 diabetes and mild to moderate renal impairment secondary to diabetic nephropathy.

Objectives:

To assess the suppressive effect of Cilostazol on the progression of diabetic nephropathy, as defined by rates of decline in glomerular filtration rate, serum creatinine and urinary albumin excretion rate.

The rising prevalence of diabetes in Asia imposes a heavy burden on the health care system. Given the increasingly early onset of disease, patients with type 2 diabetes have long duration of disease for the development of complications. Among all complications, microangiopathic complications are major causes of mortality and morbidity in diabetic patients. In Asia, patients with type 2 diabetes are particularly susceptible to the development of nephropathy. Among dialysis patients, the primary disease is diabetic nephropathy in about 40 to 50 % of patients. Despite the inhibition of the renin angiotensin system using either ACE inhibitor or AII receptor blocker (ARB) as well as introduction of tight glycaemic and blood pressure control, the prevalence of diabetic nephropathy remains high. More importantly, patients with nephropathy have more adverse metabolic profiles and increased risk of having other complications such as retinopathy, macrovascular diseases and neuropathy than those without. Indeed, according to the RENAAL Study, despite receiving the best of care, the combined event rate of death, cardiovascular disease and end stage renal disease in diabetic patients with renal impairment remained as high as 10% per year.

Cilostazol exerts antiplatelet, antithrombotic and vasodilating effects by inhibiting phosphodiesterase type 3 in platelets and vascular smooth muscle cells. Furthermore, cilostazol treatment has been shown to reduce serum triglyceride concentrations and increase HDL-cholesterol levels. In Japanese patients with type 2 diabetes, cilostazol therapy was associated with regression of carotid intimal media thickness and could prevent the onset of silent brain infarction. On the other hand, abnormal metabolism of prostaglandins in renal glomeruli has been postulated to modulate renal haemodynamics. Elevated levels of platelet-derived microparticles and soluble adhesion molecules may further contribute to the development of diabetic nephropathy. Cilostazol treatment had been shown to reduce serum levels of PMP, activated platelet subsets, soluble adhesion molecules and urinary excretion of thromboxane B2 in patients with type 2 diabetes. These changes were accompanied by a reduction in urinary albumin excretion and an increase in creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 20 and 70 years
2. Patients with Type 2 diabetic mellitus
3. A fasting urinary albumin/creatinine ratio greater than or equal to 30 mg/mmol or 24 hour urinary albumin excretion greater than or equal to 300 mg/day in two urine collections during the baseline period
4. Two consecutive serum creatinine levels during baseline period which meet the following requirements:

   * Women: between 80 umol/l and 250 umol/l (inclusive)
   * Men: between 105 umol/l and 250 umol/l (inclusive)
5. Written informed consent

Exclusion Criteria:

* Pregnancy
* Known allergy to cilostazol or aspirin
* Congestive heart failure (NYHA class III to IV)
* Severe liver impairment (greater than or equal to 3 times ULN of ALT)
* Serum potassium levels greater than or equal to 5.5 mmol/l on 2 consecutive specimens

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Doubling of serum creatinine level | 1 year
50% reduction in GFR (estimated by MDRD equation) | 1 year
GFR less than 15 ml/min/1.73m2 | 1 year
Need for dialysis | 1 year
Death related to renal causes | 1 year
Fatal or severe bleeding | 1 year

SECONDARY OUTCOMES:
Composite cardiovascular endpoints (acute myocardial infarction, revascularisation procedures, heart failure or unstable angina or arrhythmia) requiring hospital admissions, lower extremity amputation) | 1 year
Number of hospital admissions, total number of days of hospital stay and attendance at the Accident and Emergency Department | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Tong, PhD, MBBS, Principal Investigator — Chinese University of Hong Kong